CLINICAL TRIAL: NCT05649332
Title: Open, Non-comparative, Multicentre, Interventional Post-market Clinical Follow-up (PMCF) Study to Evaluate the Performance and Safety of the Medical Device Argogen® (adsorbing Spray Powder for Exudates with Silver Ions) in the Treatment of Pressure Ulcers and Minor (first and Second Degree) Burn Wounds
Brief Title: Study to Evaluate the Performance and Safety of the Medical Device Argogen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Signorini Medicale S.r.l. (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Signorini Medicale S.r.l.
Record Dates: First submitted 2022-11-16; First posted 2022-12-14 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Burn Wound; Pressure Ulcers Stage II; Pressure Ulcers Stage III
Keywords: Burn Wound; Minor Burn Wounds; Superficial Burn Wounds; Deep Partial thickness Burn Wounds; Pressure ulcers; pressure sores; bed sores; decubitus ulcers
MeSH Terms: conditions — Burns; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects presenting pressure ulcers or burn wounds (Experimental): Subjects will be treated with the medical device Argogen® adsorbing spray powder. The dosage will depend on the patient's skin condition and the extent of the areas to be treated. The medical device will be used twice a day without interruption for the duration of the study (4 weeks) or until complete healing.
  Interventions: Device: Argogen (silver zeolite powder)

INTERVENTIONS:
Device: Argogen (silver zeolite powder) — The medical device will be self-administered by each patient twice daily without interruption for the duration of the study (4 weeks) or until complete healing. Application is carried out by spraying at short intervals, lightly pressing the dispenser button and directing the spray onto the area to be treated.

SUMMARY:
A wound, i.e., a break in the skin, can result from several reasons. Pressure ulcers (also called pressure sores, bed sores and decubitus ulcers) are localized damage to the skin and underlying soft tissue usually over a bony prominence or related to a medical or other device, occurring as a result of intense and/or prolonged pressure or pressure in combination with shear.

Burn wounds result from traumatic injuries to the skin or other tissues primarily caused by heat, electrical discharge, friction, chemicals, or radiation. Burns are acute wounds caused by an isolated, non-recurring insult.

The Medical Device Argogen® (adsorbing spray powder for exudates with silver ions) consists of silver zeolite powder, combining in a single physical form the adsorbing properties of the zeolite structure and the antimicrobial properties of silver.

Its action is due to the porous structure of zeolite that actively absorbs and control wounds exudate, keeping clean and dry the environment of small skin lesions, as wounds, abrasions, minor burns and bedsores. The association with silver ions gives to the medical device the additional property of an antimicrobial effect.

The present study is to confirm that in a population of men and women presenting minor burn wounds (superficial or superficial / deep partial thickness) or chronic pressure ulcers stage 2 or 3 - NPUAP Classification (partial-thickness skin loss with exposed dermis or full-thickness skin loss) the medical device already CE marked Argogen® (adsorbing spray powder for exudates with silver ions) safely attests its capacity to promote wound healing, evaluated as percentage (%) of subjects with objective signs of wound healing (evaluated by mean of VSS score reduction for burn wounds or PUSH tool score reduction for pressure ulcers), results observed after 2 and 4 weeks after the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* In- or outpatients of both sexes, of all ethnic backgrounds, aged between 18 and 75 years(inclusive).
* Patients presenting superficial / first degree and superficial / deep partial-thickness / second degree burn wound in less than 10% of total body surface area, for which the burning event occurred within 48 hours and that can be treated within 24 hours after enrolment in the study (at baseline) or patients presenting chronic pressure ulcers stage 2 or 3 (according to the NPUAP Classification) that did not heal within 3 weeks despite proper wound care, with areas (or scattered areas) of necrosis (nonviable soft tissue/slough) more than 40%, and with a target wound which is between 4 cm squared to 20 cm squared in area at the baseline assessment.
* Patients, who are, in the opinion of the Investigator, able to understand this study, cooperate with the study procedures and are willing to return to the centre (if outpatients) for all the required visits.
* Patients who have given their written informed consent in accordance with provisions of pertinent excerpt from the Declaration of Helsinki and the Romanian laws.

Exclusion Criteria:

* Severe heart (myocardial infarction, myocardial damage, etc.), brain, liver, kidney, lung and other organ disease.
* Medical history or not-treated diabetes mellitus or diabetic foot syndrome.
* Peripheral artery disease with ankle brachial index (ABI < 0.9).
* Thrombocytopenic patients (platelet <150.000 g/l; collected in last 3 months medical history).*
* Haemoglobin < 95 g/l (collected in last 3 months medical history).*
* Concomitant infection of another site or osteomyelitis or erysipelas or phlegmon.
* Complicated deep tissue infection requiring systemic antimicrobial therapy.
* Active viral hepatitis (A/B/C) or active HIV infection or active syphilis.
* Presence of neoplastic growth in the ulcer.
* History or clinical signs of impairment of the cochlea or vestibularis system.
* Neuromuscular diseases (i.e., myasthenia gravis, Parkinson's disease)
* Aminoglycoside treatment or other antibiotic treatments for chronic venous ulcers administered less than four weeks before inclusion.
* Concomitant administration of proteolytic enzymes or products containing proteolytic enzymes (i.e., bromelain, chymotrypsin, ficin, papain, serrapeptase, trypsin) during the whole study.
* Pregnant woman, lactating woman, and man or woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception** during the study.

  **Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
* Known allergy to the tested medical device and its components (in particular, allergy to silver).
* Patients with any other medical condition that, in the opinion of the Investigator, would compromise participation or be likely to lead to hospitalisation during the study.
* Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.

  * If such lab tests are not available at screening a blood sample can be collected for analyses. However, the patient can be enrolled and start immediately treatment.

After Visit 1, the Investigator will examine the laboratory results, as soon as available, to determine patient continuation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall performance of Argogen spray® in safely promoting wound healing according to following evaluations | 2 - 4 weeks
  of pressure ulcers: percentage of subjects with objective signs of wound healing, assessed through the validated Pressure Ulcer Scale for Healing tool (PUSH ver. 3.0score) evaluated by Investigator and burn wounds: percentage (%) of subjects with objective signs of wound healing, assessed through the validated Vancouver Scar Scale (VSS), evaluated by Investigator.
To evaluate the overall safety of Argogen spray® in safely promoting wound healing according to following evaluations | 2 - 4 weeks
  Adverse Events, Serious Adverse Events, Adverse Device Events, Serious Adverse Device Events, Anticipated Serious Adverse Device Events, Unanticipated Serious Adverse Device Events incidence assessed by Investigator and reported according to the current legislation.

SECONDARY OUTCOMES:
Assessment of wound bed, wound edge, periwound skin status, performed by the Investigator | 2 - 4 weeks
  Assessment of wound bed, wound edge, periwound skin status, performed by the Investigator at 2 and 4 weeks after the initiation of treatment, compared to day 0 (baseline), based on skin appearance. The lower the percentage and affected surface - cm, the better evolution of healing compared to baseline.
Time to healing evaluated by the Investigator | 2 - 4 weeks
  The investigator will assess the time of healing
Pain assessment assessed by the Subject | 2 - 4 weeks
  Evaluation of pain due to burn wound or pressure ulcer will be done according to a Visual Analogue Scale.
  The rating will be made on 100 mm line/scale in which 0 is meaning no pain and 100 is meaning very severe pain.
  The subject has to place a vertical mark on a 100mm line to indicate how bad does he/she feels the pain at the moment of completing the questionnaire.
To assess the subject satisfaction with the treatment | 2 - 4 weeks
  The subject will assess the satisfaction with the treatment by means of the treatment satisfaction questionnaire using the four-point scale in which the subject has to place an "X" mark in the box that fits with his/ her situation:
  Very Satisfied, Satisfied, Moderately satisfied, Not satisfied.
To evaluate the global performance of Argogen | 2 - 4 weeks
  To evaluate the global performance of Argogen® by means of the Investigator Global Assessment of Performance, assessed by Investigator, through photos taken at each visit and by the performance of the treatment questionnaire using a 4-point scale:
  * 1= very good performance
  * 2 = good performance
  * 3 = moderate performance
  * 4 = poor performance
To evaluate the global safety of Argogen | 2 - 4 weeks
  To evaluate the global safety of Argogen® by means of the Investigator / Patient Global
  Assessment of Safety assessed by the Investigator and by the patient using a 4-point scale:
  * 1= very good safety
  * 2 = good safety
  * 3 = moderate safety
  * 4 = poor safety

CONTACTS AND LOCATIONS:
Overall Officials: Lorel Muresan, PhD, Principal Investigator — SC Salvosan Ciobanca SRL; Simona L Ianosi, PhD, Principal Investigator — MC Medica SRL
Locations (2):
- Romania (2):
  - MC Medica SRL, Craiova, Dolj
  - SC Salvosan Ciobanca SRL, Zalău, Sălaj County

REFERENCES:
- [Background] Sood A, Granick MS, Tomaselli NL. Wound Dressings and Comparative Effectiveness Data. Adv Wound Care (New Rochelle). 2014 Aug 1;3(8):511-529. doi: 10.1089/wound.2012.0401. PMID 25126472
- [Background] Edsberg LE, Black JM, Goldberg M, McNichol L, Moore L, Sieggreen M. Revised National Pressure Ulcer Advisory Panel Pressure Injury Staging System: Revised Pressure Injury Staging System. J Wound Ostomy Continence Nurs. 2016 Nov/Dec;43(6):585-597. doi: 10.1097/WON.0000000000000281. PMID 27749790
- [Background] Abazari M, Ghaffari A, Rashidzadeh H, Badeleh SM, Maleki Y. A Systematic Review on Classification, Identification, and Healing Process of Burn Wound Healing. Int J Low Extrem Wounds. 2022 Mar;21(1):18-30. doi: 10.1177/1534734620924857. Epub 2020 Jun 11. PMID 32524874
- [Background] Kagan RJ, Peck MD, Ahrenholz DH, Hickerson WL, Holmes J 4th, Korentager R, Kraatz J, Pollock K, Kotoski G. Surgical management of the burn wound and use of skin substitutes: an expert panel white paper. J Burn Care Res. 2013 Mar-Apr;34(2):e60-79. doi: 10.1097/BCR.0b013e31827039a6. No abstract available. PMID 23446645
- [Background] Fan K, Tang J, Escandon J, Kirsner RS. State of the art in topical wound-healing products. Plast Reconstr Surg. 2011 Jan;127 Suppl 1:44S-59S. doi: 10.1097/PRS.0b013e3181fbe275. PMID 21200273
- [Background] Atiyeh BS, Costagliola M, Hayek SN, Dibo SA. Effect of silver on burn wound infection control and healing: review of the literature. Burns. 2007 Mar;33(2):139-48. doi: 10.1016/j.burns.2006.06.010. Epub 2006 Nov 29. PMID 17137719
- [Background] Cavanagh MH, Burrell RE, Nadworny PL. Evaluating antimicrobial efficacy of new commercially available silver dressings. Int Wound J. 2010 Oct;7(5):394-405. doi: 10.1111/j.1742-481X.2010.00705.x. PMID 20626470
- [Background] Wright JB, Lam K, Hansen D, Burrell RE. Efficacy of topical silver against fungal burn wound pathogens. Am J Infect Control. 1999 Aug;27(4):344-50. doi: 10.1016/s0196-6553(99)70055-6. PMID 10433674
- [Background] Matsumura Y, Yoshikata K, Kunisaki S, Tsuchido T. Mode of bactericidal action of silver zeolite and its comparison with that of silver nitrate. Appl Environ Microbiol. 2003 Jul;69(7):4278-81. doi: 10.1128/AEM.69.7.4278-4281.2003. PMID 12839814
- [Background] Kwakye-Awuah B, Williams C, Kenward MA, Radecka I. Antimicrobial action and efficiency of silver-loaded zeolite X. J Appl Microbiol. 2008 May;104(5):1516-24. doi: 10.1111/j.1365-2672.2007.03673.x. Epub 2007 Dec 20. PMID 18179543
- [Background] Saeidinia A, Keihanian F, Lashkari AP, Lahiji HG, Mobayyen M, Heidarzade A, Golchai J. Partial-thickness burn wounds healing by topical treatment: A randomized controlled comparison between silver sulfadiazine and centiderm. Medicine (Baltimore). 2017 Mar;96(9):e6168. doi: 10.1097/MD.0000000000006168. PMID 28248871
- [Background] Passaglia E. Zeoliti naturali, zeolititi e loro applicazioni [Internet]. [cited 2022 Jun 27]. Available from: https://www.unilibro.it/libro/passaglia-elio/zeoliti-naturali-zeolititi-loro-applicazioni/9788887801194
- [Background] Rai M, Yadav A, Gade A. Silver nanoparticles as a new generation of antimicrobials. Biotechnol Adv. 2009 Jan-Feb;27(1):76-83. doi: 10.1016/j.biotechadv.2008.09.002. Epub 2008 Sep 30. PMID 18854209
- [Background] Tsipouras N, Rix CJ, Brady PH. Passage of silver ions through membrane-mimetic materials, and its relevance to treatment of burn wounds with silver sulfadiazine cream. Clin Chem. 1997 Feb;43(2):290-301. PMID 9023132
- [Background] Burd A, Kwok CH, Hung SC, Chan HS, Gu H, Lam WK, Huang L. A comparative study of the cytotoxicity of silver-based dressings in monolayer cell, tissue explant, and animal models. Wound Repair Regen. 2007 Jan-Feb;15(1):94-104. doi: 10.1111/j.1524-475X.2006.00190.x. PMID 17244325
- [Background] Luo SH, Xiao W, Wei XJ, Jia WT, Zhang CQ, Huang WH, Jin DX, Rahaman MN, Day DE. In vitro evaluation of cytotoxicity of silver-containing borate bioactive glass. J Biomed Mater Res B Appl Biomater. 2010 Nov;95(2):441-8. doi: 10.1002/jbm.b.31735. PMID 20878930
- [Background] Bondarenko O, Juganson K, Ivask A, Kasemets K, Mortimer M, Kahru A. Toxicity of Ag, CuO and ZnO nanoparticles to selected environmentally relevant test organisms and mammalian cells in vitro: a critical review. Arch Toxicol. 2013 Jul;87(7):1181-200. doi: 10.1007/s00204-013-1079-4. Epub 2013 Jun 1. PMID 23728526
- [Background] Wadhera A, Fung M. Systemic argyria associated with ingestion of colloidal silver. Dermatol Online J. 2005 Mar 1;11(1):12. No abstract available. PMID 15748553
- [Background] Pavlik V, Sojka M, Mazurova M, Velebny V. Dual role of iodine, silver, chlorhexidine and octenidine as antimicrobial and antiprotease agents. PLoS One. 2019 Jan 31;14(1):e0211055. doi: 10.1371/journal.pone.0211055. eCollection 2019. PMID 30703114
- [Background] Thomas DR, Rodeheaver GT, Bartolucci AA, Franz RA, Sussman C, Ferrell BA, Cuddigan J, Stotts NA, Maklebust J. Pressure ulcer scale for healing: derivation and validation of the PUSH tool. The PUSH Task Force. Adv Wound Care. 1997 Sep;10(5):96-101. PMID 9362591
- [Background] Stotts NA, Rodeheaver GT, Thomas DR, Frantz RA, Bartolucci AA, Sussman C, Ferrell BA, Cuddigan J, Maklebust J. An instrument to measure healing in pressure ulcers: development and validation of the pressure ulcer scale for healing (PUSH). J Gerontol A Biol Sci Med Sci. 2001 Dec;56(12):M795-9. doi: 10.1093/gerona/56.12.m795. PMID 11723157
- [Background] Chuangsuwanich A, Chortrakarnkij P, Kangwanpoom J. Cost-effectiveness analysis in comparing alginate silver dressing with silver zinc sulfadiazine cream in the treatment of pressure ulcers. Arch Plast Surg. 2013 Sep;40(5):589-96. doi: 10.5999/aps.2013.40.5.589. Epub 2013 Sep 13. PMID 24086815
- [Background] Sullivan T, Smith J, Kermode J, McIver E, Courtemanche DJ. Rating the burn scar. J Burn Care Rehabil. 1990 May-Jun;11(3):256-60. doi: 10.1097/00004630-199005000-00014. PMID 2373734
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233
- [Background] Nguyen TA, Feldstein SI, Shumaker PR, Krakowski AC. A review of scar assessment scales. Semin Cutan Med Surg. 2015 Mar;34(1):28-36. doi: 10.12788/j.sder.2015.0125. PMID 25922955
- [Background] Grey JE, Enoch S, Harding KG. Wound assessment. BMJ. 2006 Feb 4;332(7536):285-8. doi: 10.1136/bmj.332.7536.285. No abstract available. PMID 16455730
- [Background] Dowsett C, Nyløkke M. Taking wound assessment beyond the edge. Clin Pract. 2015;6(1):5.
- [Background] Inc ASI. Other Resources [Internet]. [cited 2022 Jun 27]. Available from: https://www.woundsaustralia.com.au/Web/Resources/Other_Resources/Web/Resources/Other_Resources .aspx?hkey=d5b6bb5c-78d2-4f3a-ac88-7b7f46a9afed
- [Background] CPWSC_TOWA_Brochure_210x210_No marks.pdf [Internet]. [cited 2022 Jun 27]. Available from: https://www.coloplast.com/Global/1_Corporate_website/Products/Woundcare/TOWA/CPWSC_TOWA_ Brochure_210x210_No%20marks.pdf
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Jiang ZM, Cao JD. The impact of micronized purified flavonoid fraction on the treatment of acute haemorrhoidal episodes. Curr Med Res Opin. 2006 Jun;22(6):1141-7. doi: 10.1185/030079906X104803. PMID 16846547
- [Background] Stephens TJ, Sigler ML, Herndon JH Jr, Dispensa L, Le Moigne A. A placebo-controlled, double-blind clinical trial to evaluate the efficacy of Imedeen((R)) Time Perfection((R)) for improving the appearance of photodamaged skin. Clin Cosmet Investig Dermatol. 2016 Mar 15;9:63-70. doi: 10.2147/CCID.S98787. eCollection 2016. PMID 27042135